CLINICAL TRIAL: NCT00955695
Title: A Randomized, Phase III Trial of Prophylactic Cranial Irradiation (PCI) in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) Who Are Nonprogressive on Gefitinib or Erlotinib
Brief Title: Radiation Therapy to the Brain or Observation in Preventing Brain Metastases in Patients With Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: KROG-4-2008-0276; CDR0000639096 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2010-01

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gefitinib

INTERVENTIONS:
Drug: erlotinib hydrochloride
Drug: gefitinib
Other: questionnaire administration
Procedure: quality-of-life assessment
Radiation: whole-brain radiation therapy

SUMMARY:
RATIONALE: Radiation therapy to the brain may be effective in preventing brain metastases in patients with advanced non-small cell lung cancer. It is not yet known whether radiation therapy is more effective than observation in patients with advanced non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to the brain to see how well it works compared with observation in preventing brain metastases in patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effectiveness of prophylactic cranial radiotherapy in patients with advanced non-small cell lung cancer that is responsive to gefitinib or erlotinib hydrochloride.

Secondary

* Determine the progression-free survival in patients treated with this regimen.
* Determine the overall survival in patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the psycho-neurological effects of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy regimens (first line vs second line), and disease response status (complete response or partial response vs stable disease). Patients are randomized to 1 of 2 treatment groups.

* Group 1: Patients undergo prophylactic brain radiotherapy.
* Group 2: Patients undergo observation. Patients complete quality of life (HVLT, K-ADL, EORTC QLQ-C30, and EORTC-BN20) questionnaires periodically.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Stage IIIB or IV disease
  * Must have had ≥ 8 weeks of gefitinib or erlotinib hydrochloride therapy
* At least 12 weeks of complete response or partial response since starting gefitinib or erlotinib hydrochloride

  * Stable disease allowed provided 1 of the following criteria is met:

    * EGFR mutation (exon 19 or 21)
    * Having ≥ 2 of the following 3 factors:

      * Female
      * Never smoked
      * Histologically confirmed adenocarcinoma of the lung
* No evidence of brain metastases by CT scan or MRI within the past 4 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 150,000/mm^3
* Bilirubin < 1.5 mg/dL
* Serum creatinine < 1.5 times upper limit of normal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Received 1 or 2 prior systemic chemotherapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
Time to symptomatic brain metastases

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Safety and tolerability of prophylactic cranial radiotherapy
Psycho-neurological effects of prophylactic cranial radiotherapy
Quality of life as measured by HVLT, K-ADL, EORTC QLQ-C30, and EORTC-BN20 questionnaires periodically

CONTACTS AND LOCATIONS:
Overall Officials: Chang Geol Lee, MD, Principal Investigator — Yonsei University